CLINICAL TRIAL: NCT06336811
Title: The Effects of Virtual Reality on Procedure-Related Emotional Appearance, Pain, Fear, and Anxiety During Phlebotomy in Children
Brief Title: Virtual Reality Distraction During Phlebotomy in Children
Acronym: activeVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DEU active-pasive VR
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pain, Acute; Child, Only; Anxiety and Fear
Keywords: phlebotomy; virtual reality
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Before blood collection, the "Emotional Appreance Scale for Children" was evaluated by a non-researcher nurse. Pediatric patients between the ages of 6 and 12, from whom blood would be collected, were distributed to groups according to the randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No additional intervention will be performed on the patient in the control group, and until the intervention begins, "How old are you?" Which grade are you in? What is the name of your favorite friend? Which sport do you enjoy doing more? His attention was distracted by asking questions such as.
- active Virtual reality (Experimental): The remote control of the virtual glasses will be given to the hand that will not be interfered with, and the child will start, slow down or stop the application herself. Samsung Gear Oculus Guest 2 headset allows watching virtual reality applications.
  Interventions: Device: active virtual reality distraction
- passive virtual reality (Experimental): It was said that he could watch videos by wearing virtual headset glasses during the procedure. A virtual reality application that will attract the attention of children was determined by the researchers.
  Interventions: Device: passive virtual reality distraction

INTERVENTIONS:
Device: passive virtual reality distraction — watching the application by wearing virtual glasses to the child during the phlebotomy
  Arms: passive virtual reality
Device: active virtual reality distraction — The remote control of the virtual glasses will be given to the hand, and the child will start, slow down or stop the application herself.
  Arms: active Virtual reality

SUMMARY:
This randomized controlled study was conducted to evaluate the effect of distraction methods using virtual reality on the emotional appearance, pain, fear, and anxiety associated with the procedure during phlebotomy in children aged 6-12 in a private blood collection unit.

DETAILED DESCRIPTION:
The data of the study was collected with Socio-demographic Data Collection Form, Emotional Appearance Scale for Children, Facial Expression Rating Scale, Child Anxiety Scale-State, and Child Fear Scale. Demographic data and mean scores obtained from the scales were compared between the virtual reality groups, and the control group.

ELIGIBILITY:
Inclusion Criteria:

* The child agrees to participate in the study voluntarily.
* The parent agrees to participate in the study voluntarily.
* Obtaining consent forms from the child and parent

Exclusion Criteria:

* The child has a physical and psychological deficit that will prevent him from wearing the glasses that will be placed on his head to watch virtual reality.
* Having fever (>37.5C) and severe dehydration
* The patient did not take analgesics before the intervention

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
procedure related pain | 3 minutes after the phlebotomy
  Wong-Baker FACES (WBS) Pain Rating Scale. This scale uses in children aged 3 and older to rate pain severity, ranges from 0 (very happy/no pain) to 10 (hurts worst).
anxiety | 3 minutes before and after the phlebotomy
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
fear | 3 minutes before and after the phlebotomy
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear.
emotional apperance | 3 minutes before and after the phlebotomy
  This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'. Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5. The total score is made so that the numerical value is between 5-25 by adding the points obtained for each category. Higher scale score indicates the appearance of more negative emotional behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Gulcin Ozalp, Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerceker GO, Salmal N, Bektas I. The effect of active and passive virtual reality distractions on phlebotomy-related emotional behavior, pain, anxiety, and fear in children: A randomized controlled trial. J Pediatr Nurs. 2025 Jul-Aug;83:190-198. doi: 10.1016/j.pedn.2025.05.005. Epub 2025 May 12. PMID 40359712